CLINICAL TRIAL: NCT07353515
Title: Evaluation of Peri-implant Sulcus Fluid Stress Marker Levels in Peri-implant Health and Disease
Brief Title: Peri-Implant Sulcus Fluid Stress Markers in Health and Disease
Status: Completed | Type: Observational
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Vesile Elif Toy, Assistant Professor, Inonu University
Other Study IDs: TSA-2022-3398
Record Dates: First submitted 2026-01-09; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Peri-implantitis; Peri-implant Mucositis; Peri-Implant Health
Keywords: Cortisol; Dehydroepiandrosterone; Depression; Anxiety; Peri-implantitis; Peri-implant sulcular fluid
MeSH Terms: conditions — Peri-Implantitis; Depression; Anxiety Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Peri-implant sulcus fluid samples collected for biochemical analysis of stress-related and inflammatory markers.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Peri-implant Health: Participants diagnosed with peri-implant health based on clinical and radiographic evaluation.
  Interventions: Diagnostic Test: Psychological Assessment; Diagnostic Test: Peri-implant Sulcular Fluid Biomarker Analysis; Diagnostic Test: Peri-implant Clinical Examination
- Peri-implant Mucositis: Participants diagnosed with peri-implant mucositis based on clinical criteria.
  Interventions: Diagnostic Test: Psychological Assessment; Diagnostic Test: Peri-implant Sulcular Fluid Biomarker Analysis; Diagnostic Test: Peri-implant Clinical Examination
- Peri-implantitis: Participants diagnosed with peri-implantitis based on clinical and radiographic criteria.
  Interventions: Diagnostic Test: Psychological Assessment; Diagnostic Test: Peri-implant Sulcular Fluid Biomarker Analysis; Diagnostic Test: Peri-implant Clinical Examination; Diagnostic Test: Radiographic Assessment

INTERVENTIONS:
Diagnostic Test: Psychological Assessment — Psychological status was evaluated using the Beck Depression Inventory (BDI) and the State-Trait Anxiety Inventory (STAI).
Diagnostic Test: Peri-implant Sulcular Fluid Biomarker Analysis — Peri-implant sulcular fluid samples were collected and analyzed for cortisol, dehydroepiandrosterone (DHEA), and interleukin-6 (IL-6) levels using enzyme-linked immunosorbent assay (ELISA).
Diagnostic Test: Peri-implant Clinical Examination — Clinical peri-implant parameters including plaque index, gingival index, bleeding on probing, probing depth, clinical attachment level, and keratinized tissue width were recorded using a periodontal probe.
Diagnostic Test: Radiographic Assessment — Marginal bone levels around dental implants were assessed using standardized periapical radiographs.
  Groups: Peri-implantitis

SUMMARY:
This study examines the association between psychosocial stress and peri-implant diseases. Peri-implant diseases are inflammatory conditions affecting the tissues around dental implants and may contribute to implant failure. Stress-related hormones, including cortisol and dehydroepiandrosterone (DHEA), may influence inflammatory responses in peri-implant tissues.

In this study, peri-implant sulcular fluid samples are collected from patients with peri-implant health, peri-implant mucositis, and peri-implantitis. Levels of cortisol, DHEA, and interleukin-6 (IL-6) are analyzed. Anxiety and depression levels are assessed using standardized questionnaires, and clinical peri-implant parameters are recorded.

The purpose of this study is to evaluate the relationship between stress-related biomarkers, psychological status, and peri-implant health and disease.

DETAILED DESCRIPTION:
Peri-implant diseases are inflammatory conditions affecting the soft and hard tissues surrounding dental implants and represent a major cause of implant failure. Psychosocial stress is known to influence immune function through activation of the hypothalamic-pituitary-adrenal (HPA) axis, resulting in altered secretion of stress-related hormones such as cortisol and dehydroepiandrosterone (DHEA). These hormonal changes may modulate inflammatory processes in peri-implant tissues.

This cross-sectional clinical study included 62 patients with dental implants, who were divided into three groups based on clinical and radiographic criteria: peri-implant health (PH, n=18), peri-implant mucositis (PM, n=22), and peri-implantitis (PI, n=22). Depression and anxiety levels were assessed using the Beck Depression Inventory (BDI) and the State-Trait Anxiety Inventory (STAI).

Clinical peri-implant parameters, including plaque index, gingival index, bleeding on probing, probing depth, clinical attachment level, and keratinized tissue width, were recorded. Marginal bone loss was evaluated using standardized periapical radiographs. Peri-implant sulcular fluid samples were collected and analyzed for cortisol, DHEA, and interleukin-6 (IL-6) levels using enzyme-linked immunosorbent assay (ELISA). Biomarker results were expressed as both concentration and total amount.

The study evaluates the associations between psychosocial stress markers, inflammatory biomarkers, and clinical peri-implant parameters to better understand the psychoneuroimmunological mechanisms involved in peri-implant diseases.

ELIGIBILITY:
Inclusion Criteria:

* Being volunteer to participate in the study
* Adults aged 18 to 65 years.
* Systemically healthy individuals.
* No periodontal treatment within the past 6 months.
* No self-reported psychiatric disorders.
* No use of antibiotics within the past 6 months.
* No use of steroid, immunosuppressive, or psychiatric medications.
* No clinically evident oral infection.
* Not pregnant and not breastfeeding.
* Not smoking
* Maintaining oral hygiene

Exclusion Criteria:

* Age younger than 18 years or older than 65 years.
* History of periodontal treatment within the past 6 months.
* Use of antibiotics within the past 6 months.
* Inadequate or contaminated peri-implant sulcular fluid samples.
* Pregnancy or breastfeeding.
* Long-term corticosteroid usage.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population consisted of adult individuals aged 18-65 years with at least one functional dental implant. Participants were selected from patients attending the Department of Periodontology, Faculty of Dentistry, Inonu University, and were classified into peri-implant health, peri-implant mucositis, or peri-implantitis groups based on clinical and radiographic criteria.
Sampling Method: Non-Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2023-02-15 (Actual); Primary Completion 2023-12-15 (Actual); Study Completion 2024-06-15 (Actual)

PRIMARY OUTCOMES:
Peri-implant Sulcular Fluid Cortisol Level | At baseline
  Peri-implant sulcular fluid cortisol levels were measured using enzyme-linked immunosorbent assay (ELISA). Biomarker amounts were initially calculated as ng per 30 seconds of collection time and subsequently expressed as concentrations (ng/mL) for analysis and comparison among peri-implant health, peri-implant mucositis, and peri-implantitis groups.
Peri-implant Sulcular Fluid Interleukin-6 Level | At baseline (single assessment)
  Interleukin-6 levels in peri-implant sulcular fluid were measured using enzyme-linked immunosorbent assay (ELISA). Biomarker amounts were calculated as pg per 30 seconds of collection time and subsequently expressed as concentrations (ng/mL) for analysis and comparison among peri-implant health, peri-implant mucositis, and peri-implantitis groups.
Peri-implant Sulcular Fluid DHEA Level | At baseline (single assessment)
  Peri-implant sulcular fluid dehydroepiandrosterone (DHEA) levels were measured using enzyme-linked immunosorbent assay (ELISA). Biomarker amounts were calculated as ng per 30 seconds of collection time and subsequently expressed as concentrations (ng/mL) for analysis and comparison among peri-implant health, peri-implant mucositis, and peri-implantitis groups.

SECONDARY OUTCOMES:
Anxiety Scores (State-Trait Anxiety Inventory) | At baseline (single assessment)
  Anxiety levels were assessed using the State-Trait Anxiety Inventory (STAI), which consists of two subscales: the State Anxiety scale (STAI-I) and the Trait Anxiety scale (STAI-II). Each subscale includes 20 items, with total scores ranging from 20 to 80. Higher scores indicate greater levels of anxiety.
Depression Score (Beck Depression Inventory) | At baseline
  Depression levels were assessed using the Beck Depression Inventory (BDI), a 21-item self-report questionnaire. Total scores range from 0 to 63, with higher scores indicating greater severity of depressive symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Vesile E Toy, PhD, Principal Investigator — Inonu University, Department of Periodontology Faculty of Dentistry; Furkan Kuşoğlu, DDS, Study Chair — Inonu University, Department of Periodontology Faculty of Dentistry
Locations (1):
- Inonu University, Faculty of Dentistry, Malatya, Battalgazi, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Study data will be shared upon request by primary investigator Dr Vesile Elif toy elif.toy@inonu.edu.tr